CLINICAL TRIAL: NCT02439658
Title: Genetics of QT Prolongation With Antiarrhythmics
Acronym: DOFEGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mayo Clinic (Other); The Cleveland Clinic (Other); University of Colorado, Denver (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Newton-Cheh, MD, Overall Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2013P001851; 5R01HL143070 (NIH)
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Long QT Syndrome; Drug Toxicity
Keywords: genetic research
MeSH Terms: conditions — Long QT Syndrome; Drug-Related Side Effects and Adverse Reactions | interventions — dofetilide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dofetilide patients: Patients admitted for dofetilide initiation
  Interventions: Drug: Dofetilide and/or sotalol
- Sotalol patients: Patients admitted for sotalol initiation
  Interventions: Drug: Dofetilide and/or sotalol

INTERVENTIONS:
Drug: Dofetilide and/or sotalol — This is an observational study of patients receiving Dofetilide and/or sotalol as part of their routine clinical care. Patients receiving either of these medications will be compared with population controls for genetic analysis.
  Other Names: Tikosyn

SUMMARY:
To assess the ability of common genetic variants in aggregate to predict drug-induced QT prolongation in patients being loaded with dofetilide or sotalol.

DETAILED DESCRIPTION:
This study is a multi-center study attempting to identify genetic and other factors that influence QT interval response to dofetilide or sotalol. One of the goals of this study is to determine whether genetics might identify individuals at low enough genetic risk for QT prolongation that outpatient initiation might be feasible. The dofetilide or sotalol use will be solely determined by clinical staff independent of the research study based on standard clinical care. The research components of this study include only the additional collection of blood for genetic analysis, collection of subject data on a CRF and copies of electrocardiograms performed as part of routine clinical care. This study will be overseen and coordinated at MGH. Other hospitals that may participate include Mayo Clinic, Cleveland Clinic, and University of Colorado Hospital; local IRB approval will be sought at each of these centers. Data will be collected at each individual hospital by co-investigators/site PIs and stored locally according to IRB requirements. Copies of CRFs, ECGs and blood samples for genetic analysis will be forwarded to MGH, which will serve as a coordinating and analysis center (as well as a recruiting center). Data will be encoded where possible; however, due to the impracticality of removing patient identifiers from certain data types, such as medication lists and ECGs, some data containing patient information will be transported and stored at MGH. Dr. Newton-Cheh will serve as overall study PI.

The investigators propose to conduct a research study to examine known and explore potentially unknown genetic predictors of QT response in patients being admitted for dofetilide or sotalol initiation as part of their routine clinical care. Any patient being admitted to a participating institution for the purpose of dofetilide or sotalol initiation will be eligible. Patients must be able to understand the risks of genetic testing, and be willing to undergo a venipuncture for blood collection for genotyping. Exclusion criteria include inability to provide informed consent. The investigators have a goal to enroll a total of 1000 study participants across all collaborating centers.

Patients will be identified by investigators based on planned admission for dofetilide or sotalol initiation, and following explanation of the study by co-investigator, will be asked about study participation and informed consent will be obtained. Investigators will complete a data collection form for each patient, which will include contact information, demographic information, clinical information, family history and pedigree, and all electrocardiography information available (tracings, reports). Patients will then undergo venipuncture, and two 5mL blood samples (tubes) will be collected for genotyping. Patients will also be consented for future re-contact about additional data, information, or samples needed for analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for dovetailed or sotalol initiation for clinical purposes.

Exclusion Criteria:

* Inability to provide informed consent
* Inability to provide blood samples for DNA testing (anemia, coagulopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for dovetailed or sotalol initiation for clinical purposes.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
QT interval | QT intervals will be measured on each ECG obtained during the index hospitalization
  QT interval will be measured on electrocardiograms, and recorded in the case report form

SECONDARY OUTCOMES:
Successful drug initiation | Patient will be followed for the duration of the hospitalization, which is on average 3 days
  This outcome will be recorded in the case report form

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Newton-Cheh, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - University of Colorado Hospital, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio